CLINICAL TRIAL: NCT02092428
Title: Contrast- Enhanced Whole-Heart Coronary Magnetic Resonance Angiography (MRA) at 3.0T
Brief Title: Contrast- Enhanced Whole-Heart Coronary MRA at 3.0T (Tesla)
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Cedars-Sinai Medical Center (Other)
Collaborators: National Institute for Biomedical Imaging and Bioengineering (NIBIB) (NIH)
Responsible Party: Principal Investigator, Debiao Li, PhD, Director, Biomedical Imaging Research Institute, Cedars-Sinai Medical Center
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: 23311; 5R01EB002623-07 (NIH)
Record Dates: First submitted 2014-03-04; First posted 2014-03-20 (Estimated); Last update posted 2018-03-23 (Actual); Status verified 2018-03

CONDITIONS: Coronary Artery Disease
Keywords: Coronary Magnetic Resonance Imaging; CAD; Coronary Magnetic Resonance Angiography; MRA; 3 Tesla MRI
MeSH Terms: conditions — Coronary Artery Disease | interventions — Image Enhancement; Magnetic Resonance Spectroscopy; Contrast Media; Adenosine; regadenoson

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Image Quality (Experimental): Healthy volunteers and patients will undergo non-contrast MRI or contrast-enhanced MRI to compare image quality between contrast and non-contrast scans.
  Interventions: Other: Image Quality
- Diagnostic Accuracy (Experimental): Healthy volunteers and patients will undergo non-contrast MRI or contrast-enhanced MRI to assess the diagnostic accuracy of coronary MRI in detecting CAD as compared to conventional x-ray angiography
  Interventions: Other: Diagnostic Accuracy

INTERVENTIONS:
Other: Image Quality — The following procedures may be conducted as part of this study:
  * Coronary MRI scan with no contrast
  * Coronary MRI scan enhanced with a gadolinium-based contrast agent (Optimark, MultiHance, Ablavar) administered intravenously at a total dose of up to 0.2 mmol/kg
  * MRI scan with an oral beta blocker (metoprolol)
  * Cardiac Stress Test MRI scan with a pharmacologic stress drug; either adenosine (dosage depends on the subject's weight and is set at 140mcg/kg/min) or regadenoson (0.4mg/5ml bolus)
  Determination of study drugs will be made depending upon study focus, subjects' health conditions, blood pressure, heart rate and concomitant medications. Both groups are eligible for all combinations of interventions.
  Other Names: MRI with contrast; contrast-enhance MRI; non-contrast MRI; gadolinium-based contrast; adenosine; regadenoson
  Arms: Image Quality
Other: Diagnostic Accuracy — Both groups are eligible for all combinations of interventions. This arm will also include collection of conventional x-ray angiography.
  Other Names: conventional x-ray angiography.; contrast-enhanced MRI; non-contrast MRI; gadolinium-based contrast; adenosine; regadenoson
  Arms: Diagnostic Accuracy

SUMMARY:
Investigators at the Biomedical Imaging Research Institute (BIRI) at Cedars-Sinai Medical Center have developed a Magnetic Resonance Imaging (MRI) method for imaging coronary arteries using slow-infusion, contrast-enhanced data acquisition. This method allows faster data acquisition and better spatial resolution.

Specific aims of this study are to:

1. compare coronary artery imaging with and without contrast media on both healthy subjects and patients;
2. assess the accuracy of coronary MRI in detecting coronary artery disease as compared to conventional x-ray angiography

Researchers hypothesize that contrast-enhanced MRI will improve the delineation of coronary arteries over non-contrast-enhanced MRI and that optimized, contrast-enhanced coronary MRI technique will accurately detect coronary artery disease (CAD) as compared to conventional x-ray angiography.

DETAILED DESCRIPTION:
This is a study to compare image quality between contrast and non-contrast cardiac MR and to evaluate the diagnostic accuracy of a cardiac MRI procedure in a patient population that includes both healthy volunteers and a study group of patients with known CAD who are scheduled for clinical coronary angiography within one month of signing informed consent. Both groups are eligible for a combination of imaging tests. Subjects may receive either a non-contrast MRI or a contrast-enhanced MRI depending upon their kidney function and study focus. Also based upon the focus of the study at the time of the scan and to improve image quality, a beta-blocker to lessen motion artifact in patients with higher heart rates may be administered or patients may be asked to undergo a stress test for comparison.This is a one-day research procedure. Studies are acquired from the approved Institutional Review Board #25881 Cedars-Sinai Biomedical Imaging Research Registry.

ELIGIBILITY:
Inclusion:

* All subjects must be enrolled in the IRB approved Cedars-Sinai Biomedical Imaging Research Registry where data is collected for this analysis study.
* Male or female ≥ 18years of age
* Healthy Group -No known CAD
* CAD Group-Scheduled for clinical invasive coronary artery x-ray angiography within one month of study participation

Exclusion:

* MR imaging is contraindicated in persons with mechanically, magnetically, or electrically activated implants, such as cardiac pacemakers, neurostimulators, and infusion pumps.
* Persons with ferromagnetic implants and ferromagnetic foreign bodies, such as intracranial, aneurysm clips, shrapnel and intraocular metal chips as these could become dislodged.
* Patients who are pregnant, nursing are implanted with intrauterine devices (IUD's)
* Persons who are in atrial fibrillation at the time of the MR scan as this could result in poor image quality due to interference with electrocardiographic gating necessary for image acquisition.
* Persons unable to tolerate MRI imaging secondary to an inability to lie supine or severe claustrophobia.
* Patient with renal failure (GFR< 45)
* Allergy to animal dander or animal-instigated asthma
* Specific to Ablavar: Baseline ECG measurements and concomitant medications will be checked on subjects who are chosen to participate in the Ablavar study, based upon study needs. If the ECG measurements and/or medications indicate that the subject is at high risk for arrhythmia, the subject will be excluded from the Ablavar study, but can participate in the OptiMark/MultiHance contrast study or non-contrast study.
* Specific to beta-blocker administration: no contraindication to beta blockers. If the subject is found to have a contraindication to beta-blockers or declines the administration of beta-blockers the subject will be excluded from the beta-blocker portion but can still participate in a non-contrast or contrast-enhanced scan without beta-blocker administration.
* Specific to Regadenoson: no contraindication to regadenoson administration. If the subject is found to have a contraindication to regadenoson the subject will be excluded from the regadenoson portion but can still participate in a non-contrast or contrast-enhanced scan without regadenoson stress testing.
* Specific to Adenosine: no contraindication to adenosine administration.If the subject is found to have a contraindication to adenosine the subject will be excluded from the adenosine portion but can still participate in a non-contrast or contrast-enhanced scan without adenosine stress testing.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 333 (Actual)
Dates: Start 2011-04 (Actual); Primary Completion 2017-03-01 (Actual); Study Completion 2017-03-01 (Actual)

PRIMARY OUTCOMES:
Diagnostic performance of 3.0-T contrast-enhanced whole-heart coronary MRA in patients with suspected coronary artery disease (CAD) | one day
  sensitivity and specificity

CONTACTS AND LOCATIONS:
Overall Officials: Debiao Li, PhD, Principal Investigator — Cedars-Sinai Medical Center
Locations (1):
- Cedars-Sinai Medical Center, Los Angeles, California, United States